CLINICAL TRIAL: NCT03890783
Title: Evaluation of Functional Results After Surgery of Oropharyngeal Cancers With Soft Palate With Free Flap Reconstruction
Brief Title: Functional Results of Soft Palate Free Flap Reconstruction
Acronym: RECaVoLL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0826; 2018-A03408-47 (Other: ID-RCB)
Record Dates: First submitted 2019-01-30; First posted 2019-03-26 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Oropharyngeal Cancer; Palate Free Flap Reconstruction
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after surgery of oropharyngeal cancers: Patients after surgery of oropharyngeal cancers with soft palate with free flap reconstruction and adjuvant radiotherapy
  Interventions: Other: Evaluation of phonation quality; Other: Evaluation of swallowing quality; Other: global quality of life questionnaire

INTERVENTIONS:
Other: Evaluation of phonation quality — Evaluation of phonation quality by :
  * Self-evaluation: completion of the Voice Handicap Index questionnaire, in its 30 items version
  * Hetero-evaluation: reading and recording of 2 texts, and notation by 3 practitioners using the grade, rough, breathy, asthenic, strained (GRBAS) scale, to evaluate the occurrence and the gravity of rhinolalia
Other: Evaluation of swallowing quality — Evaluation of swallowing quality by:
  * Self-evaluation: completion of the Deglutition Handicap Index questionnaire
  * Hetero-evaluation: nasofibroscopy to evaluate the occurrence of aspiration and nasal regurgitation
Other: global quality of life questionnaire — Completion of the European Organization for Research and Treatment of Cancer Quality of Life questionnaire (EORTC QLQ - C30) and the EORTC QLQ - H&N35 questionnaires

SUMMARY:
The oropharynx is a complex anatomical structure necessary for nasal breathing, swallowing and phonation. The removal of oropharyngeal cancers can lead to sequelae, particularly in the case of resections affecting the soft palate. The main sequelae are represented by rhinolalia and swallowing disorders with nasal regurgitation.

The treatment of oropharyngeal tumors is based on primary surgery or radiotherapy, but tumors of the soft palate are often treated by radiotherapy or radio-chemotherapy first. Surgery is often kept for relapses, because it is considered to lead to important sequelae. However, chemoradiotherapy of the oropharynx is also responsible for acute toxicities, and late sequelae can be frequent and important.

Recent publications tend to show that primary surgery would give better survival rates compared to radiotherapy, particularly in advanced stages, including viro-induced cancers. In addition, primary surgery can reduce the dose of radiation delivered to the oropharynx and thus reduce its long-term toxicity.

It is currently possible to reconstruct a loss of substance after surgery of oropharyngeal cancers, including the soft palate by using free flaps, limiting the postoperative sequelae usually observed without reconstruction.

There is little data on reconstructions of the soft palate, their sequelae and their impact on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oropharyngeal tumor who had surgical management with removal of all or part of the soft palate and free flap reconstruction, and at least 12 month after the end of external radiotherapy treatment
* Patients over 18 years old

Exclusion Criteria:

* Patients protected by law (guardianship, curatorship and under judicial protection)
* Patients who expressed their opposition to participate to the study
* Patients who do not speak French (incompatible with reading, understanding and filling out the questionnaires)
* Patients participating in interventional research (excluding physiological studies and interventional research with minimal risks and constraints that do not interfere with the primary endpoint analysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, with oropharyngeal tumor requiring surgical management with excision of part or all of the soft palate, with free flap reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of phonation quality at least 12 months after the end of external radiotherapy. | 12 months
  Self-evaluation by completion of the Voice Handicap Index questionnaire, in its 30 items version.
  For self evaluation of phonation using the Voice Handicap Index 30 (VHI 30) questionnaire:
  The VHI is rated on 120 points. For each question a score from 0 to 4 is assigned (0 = never, 1 = almost never, 2 = sometimes, 3 = almost always, 4 = always). Its three sub-scales allow to establish an emotional score E out of 40, a physical score P out of 40 and a Functional score F out of 40.
  The total score can therefore be between 0 and 120 points. The interpretation of this test is done by comparing the sub-scores and the total score obtained with the averages values of these sub-scores and total score.

SECONDARY OUTCOMES:
Hetero evaluation of phonation quality at least 12 months after the end of external radiotherapy | 12 months
  Hetero-evaluation performed by 3 practitioners, using the Grade Roughness Breathiness Asthenia Strain (GRBAS) score, after the patient has read and recorded two texts.
  GRBAS means: G for Grade (degree of hoarseness of the voice), R for Roughness (impression of irregularity of the vibration of the vocal folds), B for Breathiness (degree to which air escaping from between the vocal folds can be heard by the examiner), A for Asthenia (degree of weakness heard in the voice), S for Strain ( extent to which strain or hyperfunctional use of phonation is heard), I for Instability (changes in voice quality over time). Each of the five parameters is rated from 0 to 3 points (0 = Normal, 1 = slightly altered, 2 = moderately impaired, 3 = severely impaired), resulting in an overall score ranging from 0 to 15. A score at 0 reflects a phonation considered normal, a score between 1 and 5 a slightly altered phonation, between 5 and 10 moderately altered and between 10 and 15 severely impaired.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Lyon Nord - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No